CLINICAL TRIAL: NCT04622527
Title: Acceptability of Virtual Reality Experience by Health Care Providers for Improving Focus and Reducing Anxiety: A Pilot Trial
Brief Title: A Study to Assess Virtual Reality by Healthcare Providers: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Relay Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Ivana T Croghan, PhD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 20-009579
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; Burn Out
Keywords: anxiety; burnout
MeSH Terms: conditions — Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Participants viewed/were exposed to all 4 paradigms but in different sequence according to the randomization. With 4 paradigms there are a total of 24 ordering sequences. With a sample of N=24, each subject was randomized to one of these 24 sequences with each subject having a unique sequence.
Who Masked: Participant
Masking Description: Virtual Reality headgear and corresponding non-Virtual Reality are pre-programmed with paradigms. Participants were unaware of the order of the experience they will view.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A = Virtual Reality paradigm A (Active Comparator): Begin with Paradigm A virtual reality headgear
  Interventions: Other: Random assigned paradigm viewing order
- B = Virtual Reality paradigm B (Active Comparator): Begin with Paradigm B virtual reality headgear
  Interventions: Other: Random assigned paradigm viewing order
- C = Non-Virtual Reality paradigm A (Sham Comparator): Begin with Paradigm A without virtual reality headgear
  Interventions: Other: Random assigned paradigm viewing order
- D = Non-Virtual Reality paradigm B (Sham Comparator): Begin with Paradigm B without virtual reality headgear
  Interventions: Other: Random assigned paradigm viewing order

INTERVENTIONS:
Other: Random assigned paradigm viewing order — Participants experience the paradigm in a random order

SUMMARY:
The purpose of this study is to evaluate the acceptability of using Virtual Reality intervention to help reduce anxiety and burnout symptoms and improve focus in the workplace.

DETAILED DESCRIPTION:
The proposed investigation will apply two novel paradigms using proprietary Virtual Reality interventions designed to reduce anxiety and inattention. We will explore whether this intervention is safe and acceptable, and whether it can impact the stress, anxiety, and difficulty in focus of employees in the workplace. Participants will view two different nature videos in two different formats. Each video will be experienced through Virtual Reality or non- Virtual Reality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of consent.
* Healthcare Professional with the Mayo Clinic.
* Not pregnant by participant self-report at time of consent.
* Have the ability to provide informed consent.
* Have no contraindicated comorbid health conditions as determined by the clinical investigators.

Exclusion Criteria:

* Currently (within the past 3 weeks) practicing mindfulness training on a weekly/regular basis.
* Currently (within the past 3 weeks) undergoing an additional program (e.g., Complementary and Alternative Medicine [CAM]) to improve quality of life.
* Currently (within 3 weeks) enrolled in another clinical or research program (e.g., CAM) which impacts the patients' quality of life (QOL), stress or anxiety.
* Currently has photosensitivity.
* Cannot tolerate virtual reality experiences.
* An unstable medical or mental health condition as determined by the physician investigator (e.g., pre-existing eye strain, seizures, dizziness, nausea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Principal Investigator — Mayo Clinic; Brent Bauer, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Croghan IT, Hurt RT, Aakre CA, Fokken SC, Fischer KM, Lindeen SA, Schroeder DR, Ganesh R, Ghosh K, Bauer BA. Virtual Reality for Health Care Professionals During a Pandemic: A Pilot Program. J Prim Care Community Health. 2022 Jan-Dec;13:21501319221086716. doi: 10.1177/21501319221086716. PMID 35352605

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a total of 4 treatment interventions to which every participant was exposed. Subjects were randomized to one of the 24 unique treatment sequences.
Groups:
- A = First Viewing of Virtual Reality Paradigm A: Paradigm A with virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigms in a random order beginning with viewing paradigm A with Virtual Reality headgear.
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- B = First Viewing of Virtual Reality Paradigm B: Paradigm B with virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigms in a random order viewing paradigm B with Virtual Reality headgear.
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- C = First Viewing of Non-Virtual Reality Paradigm A: Paradigm A without virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigms in a random order beginning with viewing paradigm A with Computer screen.
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- D = First Viewing of Non-Virtual Reality Paradigm B: Paradigm B without virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigm in a random order beginning with viewing paradigm B with Computer screen.
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
Period: Overall Study
Arm/Group | A = First Viewing of Virtual Reality Paradigm A | B = First Viewing of Virtual Reality Paradigm B | C = First Viewing of Non-Virtual Reality Paradigm A | D = First Viewing of Non-Virtual Reality Paradigm B
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A = First Viewing of Virtual Reality Paradigm A: Begin with Paradigm A virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigms in a random order beginning with Paradigm A with virtual reality headgear
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- B = First Viewing of Virtual Reality Paradigm B: Begin with Paradigm B virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigms in a random order beginning with Paradigm B with virtual reality headgear
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- C = First Viewing of Non-Virtual Reality Paradigm A: Begin with Paradigm A without virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigms in a random order beginning with Paradigm A through computer screen
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- D = First Viewing of Non-Virtual Reality Paradigm B: Begin with Paradigm B without virtual reality headgear
  Random assigned paradigm viewing order: Participants experience all 4 paradigm in a random order beginning with Paradigm B through computer screen
  The 4 paradigms are:
  A = Virtual Reality Paradigm A, B = Virtual Reality Paradigm B, C = Non-Virtual Reality Paradigm A, D = Non-Virtual Reality Paradigm B
- Total: Total of all reporting groups
Arm/Group | A = First Viewing of Virtual Reality Paradigm A | B = First Viewing of Virtual Reality Paradigm B | C = First Viewing of Non-Virtual Reality Paradigm A | D = First Viewing of Non-Virtual Reality Paradigm B | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (7.7) | 42.6 (5.2) | 49.0 (15.2) | 45.7 (12.5) | 46.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 3 | 10
  Male | 2 | 4 | 5 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 5 | 5 | 4 | 16
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anxiety Inventory (STAI Y1)
Description: STAI Y1 anxiety measurement of the change from post-test score to pre-test score.
  The STAI Y1 has 20 questions on a scale from 1 to 4. The minimum score is 20 and the maximum is 80. The lower the score the better the outcome. Our outcome looks at the difference between the post-test from the pre-test, so the minimum change score is -60 and the maximum change score is 60. A higher change in score would mean that a subject experienced a worse outcome after the paradigm, while a lower change in score shows a better outcome after the paradigm than before.
Time Frame: 2 weeks
Population: All 24 subjects experienced each of the 4 virtual reality paradigms. Before and after each paradigm, a STAI Y1 survey was given. The outcomes below shows the change between post and pre for all subjects, no matter what order they viewed the paradigm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- A = Virtual Reality Paradigm A: Paradigm A with virtual reality headgear
  Random assigned paradigm viewing order: Participants experience the paradigm in a random order
- B = Virtual Reality Paradigm B: Paradigm B with virtual reality headgear
  Random assigned paradigm viewing order: Participants experience the paradigm in a random order
- C = Non-Virtual Reality Paradigm A: Paradigm A without virtual reality headgear
  Random assigned paradigm viewing order: Participants experience the paradigm in a random order
- D = Non-Virtual Reality Paradigm B: Paradigm B without virtual reality headgear
  Random assigned paradigm viewing order: Participants experience the paradigm in a random order
Arm/Group | A = Virtual Reality Paradigm A | B = Virtual Reality Paradigm B | C = Non-Virtual Reality Paradigm A | D = Non-Virtual Reality Paradigm B
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -6.4 (5.98) | -5.8 (9.29) | -4.1 (6.22) | -5.0 (6.89)

2. Secondary Outcome: Was the Study Worthwhile
Description: Acceptability of Virtual Reality measured by a question from the satisfaction survey done at the end of the study. The question asked was "Was it worthwhile for you to participate in this research study?".
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A = Virtual Reality Paradigm A | B = Virtual Reality Paradigm B | C = Non-Virtual Reality Paradigm A | D = Non-Virtual Reality Paradigm B
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  No | 0 | 0 | 1 | 0
  Yes | 6 | 6 | 5 | 5
  Unsure | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 weeks of study participation
Arm/Group | A = Virtual Reality Paradigm A | B = Virtual Reality Paradigm B | C = Non-Virtual Reality Paradigm A | D = Non-Virtual Reality Paradigm B
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04622527/Prot_SAP_000.pdf